CLINICAL TRIAL: NCT07128888
Title: A Study to Evaluate the Effect of GZR18 Injection on Gastric Emptying and Its Drug-Drug Interactions With Digoxin, Rosuvastatin Calcium and Warfarin Sodium in Obese or Overweight Subjects
Brief Title: Study on Gastric Emptying Effect and Drug-Drug Interactions of GZR18 Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZR18-BWM-104
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Obesity or Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Rosuvastatin Calcium; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GZR18 injection (Experimental)
  Interventions: Drug: GZR18 injection,digoxin tablets, rosuvastatin calcium tablets and warfarin sodium tablets

INTERVENTIONS:
Drug: GZR18 injection,digoxin tablets, rosuvastatin calcium tablets and warfarin sodium tablets — GZR18 injection: 3 mg-36 mg，16 weeks; Warfarin Sodium Tablets:2.5mg，twice; Rosuvastatin Calcium Tablets：10mg，twice; Digoxin Tablets:0.25mg，twice

SUMMARY:
This is a single-center, open-label, fixed-sequence phase I clinical study to evaluate the effect of GZR18 Injection on gastric emptying and the effect of repeated SC injections of GZR18 Injection on the pharmacokinetics of oral digoxin tablets, rosuvastatin calcium tablets and warfarin sodium tablets.

A total of 60 obese or overweight subjects are planned to be enrolled, with no less than one-quarter of the subjects from either gender.

The study duration for each subject in this study is approximately 26 weeks: including a screening period of up to 4 weeks (W-28 to D-1), single-drug administration and dose escalation stages of 16 weeks (W1D1 to W16D7) and the combined drug administration stage of 6 weeks (W17D1 to W23D1)

ELIGIBILITY:
Inclusion Criteria:

* 1.Obese Chinese subjects, who voluntarily sign the Informed Consent Form (ICF), can receive SC injection, fully understand the content, process and possible adverse reactions of the trial, and are able to follow the regulations on contraindications and restrictions specified in this protocol.

  2. Male or female, 18 to 50 years of age at signing the ICF (both inclusive).

  3. Body mass index (BMI) within 26-35 kg/m2 (both ends inclusive) at screening.

  4. No abnormality or not clinically significant abnormality as judged by the investigator in physical examination, vital signs, routine laboratory tests (hematology, blood chemistry, urinalysis, thyroid function and coagulation), 12-lead ECG, ultrasonography of liver, gallbladder, pancreas, and spleen + both kidneys, chest imaging examination and other results. (abnormal indicators related to obesity or overweight, and the investigator assesses that they have no impact on this study, they can be enrolled)

  5. Subjects of childbearing potential with no birth plan from the signing of the ICF to 8 weeks after the last dose, willingness to take effective contraceptive measures, and no plan for sperm or ovum donation. Females of childbearing potential must not be lactating and must have negative results for blood pregnancy test at screening (including D-1).

Exclusion Criteria:

* 1.Subjects with a previous or existing history of heart, liver, kidney, gastrointestinal tract, respiratory system, nervous system, psychiatric disorders, endocrine diseases (except obesity), malignant tumors and other diseases that are judged by the investigator to have an impact on the evaluation of the results of this study.

  2. History or existing diseases that increase the risk of subjects, such as hypoglycemia, acute or chronic pancreatitis, pancreatic injury, history of symptomatic gallbladder disease; cholelithiasis with high risk of acute biliary pancreatitis at screening (e.g., silt-like lithiasis, gallbladder or bile duct stone ≤ 5 mm in diameter)，newly diagnosed cholecystitis at screening.

  3. Subjects with previous or existing clinically significant digestive system diseases who are judged unsuitable for the study by the investigator, such as history of active peptic ulcer or hemorrhage, inflammatory bowel disease, abnormal gastric emptying (such as gastric paresis or pyloric stenosis, gastric outlet obstruction), continuous use of drugs affecting gastrointestinal motility for ≥ 1 week (including but not limited to domperidone, mosapride, macrolides), and acute hemorrhoidal attacks within the past three months.

  4. History or family history of previous or existing medullary thyroid carcinoma, multiple endocrine neoplasia type 2.

  5. Subjects who have used any drugs that alter the activity of drug metabolizing enzymes or transporters within 4 weeks prior to screening, or subjects with acute diseases or concomitant medication from the screening period to before administration of the investigational medicinal product (IMP).

  6. Subjects with severe infection or unexplained infection within 4 weeks before screening.

  7. Major surgery within 6 months prior to screening, or scheduled surgery or hospitalization during the study.

  8. Subjects with allergic constitution prior to screening, or a history of bronchial asthma, eczema and other allergic diseases (except mild seasonal allergy), or a history of severe food allergy (such as laryngeal edema, shock), or known allergy to any ingredient in investigational medicinal products (IMPs) [GLP-1 receptor (GLP-1R) agonist, paracetamol, digoxin, rosuvastatin, warfarin and their excipients].

  9. Use of any prescription drugs, over-the-counter drugs or Chinese herbal medicines within 2 weeks prior to screening; or use of any GLP-1R agonists or drugs with the same mechanism of action to GLP-1R agonists [such as GLP-1R/glucagon receptor (GCGR) agonists or gastric inhibitory polypeptide receptor (GIPR)/GLP-1R agonists or GIPR/GLP-1R/GCGR agonists] within 6 months prior to screening; or use of any weight loss drugs within 6 months prior to screening.

  10. Subjects who have been vaccinated within 1 month before screening or are scheduled for vaccination during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Cmax:Maximum plasma concentration | through study completion,up to 16 weeks
AUC0-last:Area under the plasma concentration-time curve at 0 h to last observation time-point after a single dose. | through study completion,up to 16 weeks
AUC0-inf:Area under the plasma concentration-time curve at 0 h to infinity after a single dose. | through study completion,up to 16 weeks

SECONDARY OUTCOMES:
Tmax:Time of Maximum Drug Concentration | through study completion,up to 16 weeks
t1/2: Elimination half-life | through study completion,up to 16 weeks
CL/F: Apparent clearance rate | through study completion,up to 16 weeks
Vz/F:Apparent Volume of Distribution associated with the Terminal Phase following Oral Administration | through study completion,up to 16 weeks
PD:Area under the international normalized ratio-time curve (INRAUC) and maximum international normalized ratio postdose (INRMAX) for warfarin | through study completion,up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Study site 01, Beijing, China